CLINICAL TRIAL: NCT03808311
Title: Blood Pressure Control Target in Diabetes (BPROAD): a Multicenter, Open-label, Parallel-group, Randomized Controlled Trial
Brief Title: Blood Pressure Control Target in Diabetes
Acronym: BPROAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Guang Ning, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ruijin-2018-138-2
Record Dates: First submitted 2018-12-16; First posted 2019-01-17 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-08

CONDITIONS: Blood Pressure Control Target in Diabetes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intensive BP treatment arm (Experimental): Participants in the intensive BP treatment arm will be treated to a systolic BP target of <120 mmHg.
  Interventions: Other: Treatment strategy regarding different systolic BP goals
- Standard BP treatment arm (Other): Participants in the standard BP treatment arm will be treated to a systolic BP target of <140 mmHg.
  Interventions: Other: Treatment strategy regarding different systolic BP goals

INTERVENTIONS:
Other: Treatment strategy regarding different systolic BP goals — The trial will test a treatment strategy question regarding different systolic BP goals and not test specific medications. Therefore, the BP treatment protocol is flexible in terms of the choice and doses of anti-hypertensive medications as long as systolic BP levels are within targets (<120 mmHg in the intensive arm and <140 mmHg in the standard arm).

SUMMARY:
This is a multicenter, open-label, parallel-group, randomized controlled trial that will be conducted across mainland China. This trial will test the primary hypothesis of whether an intensive treatment strategy (a systolic blood pressure target of <120 mmHg) is more effective than a standard treatment strategy (a systolic blood pressure target of <140 mmHg) in reducing the risk of major cardiovascular disease (non-fatal stroke, non-fatal myocardial infarction, treated or hospitalized heart failure, and cardiovascular deaths) over a follow-up period of up to 5 years among patients with a history of diabetes and elevated systolic blood pressure. The secondary hypotheses are to compare the intensive blood pressure treatment strategy with the standard treatment strategy on cognitive function, individual components of the primary hypothesis, all-cause mortality, kidney outcomes, quality of life, and injurious falls, et al.

DETAILED DESCRIPTION:
The trial will recruit 12,702 patients from approximately 150 hospitals within the China Diabetes Clinical Research Network. Eligible criteria include men and women aged ≥50 years; type 2 diabetes mellitus; elevated systolic blood pressure; and a history of clinical cardiovascular disease or increased risk for cardiovascular disease. Main exclusion criteria include known secondary cause of hypertension, symptomatic heart failure, end-stage renal disease, and other serious illness. The proposed trial has 90% statistical power to detect a 20% reduction (hazard ratio of 0.80) in major cardiovascular disease between intensive and standard treatment groups at a 2-sided significance level of 0.05.

To achieve the proposed study objectives, the following specific aims will be accomplished:

1. Recruit 12,702 study participants who meet the eligibility criteria and randomly assign 6,351 to the intensive blood pressure treatment and 6,351 to the standard blood pressure treatment groups;
2. Achieve and maintain two-level targets of systolic blood pressure (<120 mmHg vs. <140 mmHg) with a mean systolic blood pressure difference of ≥15 mmHg;
3. Employ a study-wide strategy to encourage standard of care for all participants for the treatment of type 2 diabetes and dyslipidemia other than blood pressure;
4. Obtain clinical data on study outcomes for up to 60 months of follow-up among all trial participants;
5. Perform strict quality control procedures for intervention and data collection;
6. Conduct data analysis according to the intention-to-treat principle; and
7. Disseminate the study findings to influence clinical practice and clinical guidelines.

Findings from this trial will provide evidence as to whether intensive blood pressure management to achieve a systolic blood pressure target of <120 mmHg has additional benefits over standard management of systolic blood pressure <140 mmHg. These findings will help in the development of clinical guidelines for blood pressure management among patients with type 2 diabetes and will have important clinical impact.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged ≥50 years;
2. Diabetes defined as:

   * A self-reported previous diagnosis by health care professionals and taking anti-diabetic medications;
   * Fasting plasma glucose level of ≥126 mg/dL (7.0 mmol/L). Fasting is defined as no caloric intake for at least 8 hours;
   * 2-hour plasma glucose level of ≥200 mg/dL (11.1 mmol/L) during an oral glucose tolerance test. The test should be performed using a glucose load containing the equivalent of 75 g anhydrous glucose dissolved in water; or
   * HbA1c concentration of ≥6.5% (48 mmol/mol);
3. Systolic blood pressure

   -≥140 mmHg on 0 medication;
   * 130-180 mmHg on 1 medication;
   * 130-170 mmHg on up to 2 medications;
   * 130-160 mmHg on up to 3 medications; or
   * 130-150 mmHg on up to 4 medications;
4. Increased risk of cardiovascular disease (one or more of the following):

   * Previous history of clinical CVD (≥ 3 months)
   * Subclinical CVD within 3 years
   * 2 or more CVD risk factors
   * Estimated glomerular filtration rate (eGFR) 30-59 ml/min/1.73 m2

Exclusion Criteria:

1. History consistent with type 1 diabetes
2. Known secondary cause of hypertension
3. One minute standing systolic BP <110 mmHg
4. Arm circumference too large to allow accurate blood pressure measurement with available devices
5. Cardiovascular event or procedure or hospitalization for unstable angina within the past 3 months
6. Symptomatic heart failure within the past 6 months or left ventricular ejection fraction (by any method) <35% within the past 6 months
7. ALT or AST levels more than twice the upper limit of the normal range or active liver diseases
8. Dialysis, kidney transplantation, eGFR <30 ml/min/1.73 m2, or serum creatinine >2.0 mg/dl
9. Proteinuria
10. Previous diagnosis of polycystic kidney disease or glomerulonephritis
11. A medical condition likely to limit survival to less than 5 years
12. Any factors judged by the clinic team to be likely to limit adherence to interventions
13. Failure to obtain informed consent from participant
14. Currently participating in another intervention study
15. Currently living with another BPROAD participant
16. Pregnancy, currently trying to become pregnant, or of child-bearing potential and not using birth control

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12821 (Actual)
Dates: Start 2019-02-24 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Major cardiovascular events | 5 years
  Time to the first occurrence of any of the following: non-fatal stroke, non-fatal myocardial infarction, hospitalized or treated heart failure, or cardiovascular deaths

SECONDARY OUTCOMES:
A composite of the primary outcome and all-cause mortality | 5 years
  Time to the first occurrence of any of the following: non-fatal stroke, non-fatal MI, hospitalized or treated heart failure, or death
Macrovascular outcome | 5 years
  Time to the first occurrence of any of the following: non-fatal stroke, non-fatal MI, hospitalized or treated heart failure, cardiovascular deaths, hospitalized unstable angina, or any cardiovascular revascularization procedures
Major coronary artery diseases | 5 years
  Time to the first occurrence of any of the following: non-fatal MI, hospitalized unstable angina, revascularization of coronary arteries, or deaths due to coronary artery diseases
Total MI | 5 years
  Fatal and non-fatal MI
Total stroke | 5 years
  Fatal and non-fatal stroke
Ischemic stroke | 5 years
  Fatal and non-fatal ischemic stroke
Hemorrhagic stoke | 5 years
  Fatal and non-fatal hemorrhagic stoke
Heart failure | 5 years
  Hospitalized or treated heart failure, or heart failure death
Cardiovascular death | 5 years
  Deaths due to cardiovascular causes
Total mortality | 5 years
  Deaths due to any causes
Cognitive function | 5 years
  Time to the first occurrence of any of the following: all-cause dementia or mild cognitive impairment (MCI); all-cause dementia; MCI; changes in global cognitive function and in five specific cognitive domains
Health related quality of life | 5 years
  Evaluated with HQoL scales such as Short Form 12 Health Survey Questionnaire
Kidney outcomes | 5 years
  Progression of CKD, development of CKD, and incident albuminuria

OTHER OUTCOMES:
All cardiovascular revascularization procedures | 5 years
Hospitalized unstable angina | 5 years
Retinopathy | 5 years
Transient ischemic attack (TIA) | 5 years
Left ventricular hypertrophy (LVH) | 5 years
Atrial fibrillation or flutter | 5 years
All cancers | 5 years
  Time to the first occurrence of any types of cancer
Cost-effectiveness | 5 years
  The incremental cost per quality adjusted life year (QALY) gained. QALYs will be measured by the EuroQol-5 Dimensions (EQ-5D) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Guang Ning, MD, PhD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Ruijin hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bi Y, Li M, Liu Y, Li T, Lu J, Duan P, Xu F, Dong Q, Wang A, Wang T, Zheng R, Chen Y, Xu M, Wang X, Zhang X, Niu Y, Kang Z, Lu C, Wang J, Qiu X, Wang A, Wu S, Niu J, Wang J, Zhao Z, Pan H, Yang X, Niu X, Pang S, Zhang X, Dai Y, Wan Q, Chen S, Zheng Q, Dai S, Deng J, Liu L, Wang G, Zhu H, Tang W, Liu H, Guo Z, Ning G, He J, Xu Y, Wang W; BPROAD Research Group. Intensive Blood-Pressure Control in Patients with Type 2 Diabetes. N Engl J Med. 2025 Mar 27;392(12):1155-1167. doi: 10.1056/NEJMoa2412006. Epub 2024 Nov 16. PMID 39555827
- [Derived] Saiz LC, Gorricho J, Garjon J, Celaya MC, Erviti J, Leache L. Blood pressure targets for the treatment of people with hypertension and cardiovascular disease. Cochrane Database Syst Rev. 2022 Nov 18;11(11):CD010315. doi: 10.1002/14651858.CD010315.pub5. PMID 36398903
- [Derived] Saiz LC, Gorricho J, Garjon J, Celaya MC, Erviti J, Leache L. Blood pressure targets for the treatment of people with hypertension and cardiovascular disease. Cochrane Database Syst Rev. 2020 Sep 9;9(9):CD010315. doi: 10.1002/14651858.CD010315.pub4. PMID 32905623